CLINICAL TRIAL: NCT04847609
Title: Multicentric Observational Study of Pain When Using the GentleCath™ Air Catheter in Female Patients Followed at Home With Neurological Vesico-sphincter Disorders With Urinary Self-catheterization as a Bladder Emptying Method
Brief Title: GentleCath Air (Urinary Self-catheterization) - Pain in Female Patients With Neurological Vesico-sphincter Disorders
Acronym: FollowAir
Status: Withdrawn | Type: Observational
Why Stopped: Issues with patient recruitment
Sponsor: ConvaTec Inc. (Industry)
Collaborators: ClinSearch (Other)
Responsible Party: Sponsor
Other Study IDs: CC-20-402
Record Dates: First submitted 2021-04-01; First posted 2021-04-19 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injuries; Multiple Sclerosis; Parkinsonian Disorders; Allodynia
Keywords: Neurogenic Bladder; Intermittent Urethral Catheterization; Pain; Tolerance
MeSH Terms: conditions — Spinal Cord Injuries; Multiple Sclerosis; Parkinsonian Disorders; Hyperalgesia; Urinary Bladder, Neurogenic; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: GentleCath™ Air catheter — Patients

SUMMARY:
The purpose of this study is to evaluate the rate of occurrence of urethral pain in female patients with neurological vesico-sphincter disorders whilst performing self-catheterization using GentleCath™ Air catheters.

DETAILED DESCRIPTION:
Intermittent catheterisation involves the insertion and removal of a hollow flexible tube called a catheter to drain urine from the bladder. Intermittent catheterisation allows the individual to empty their bladder without the need for a long term indwelling catheter and can be implemented for people who have difficulty emptying their bladder due to neurogenic disorders.

One of the complaints of female patients performing intermittent self-catheterization for neurological bladder is the occurrence of urethral pain on insertion or removal of the catheter, in particular in patients retaining sensitivity at this level.

The GentleCath™ Air catheter was designed to improve its tolerance and in particular to reduce the risk of pain. However, no studies have addressed this in real life. Therefore, the purpose of this study is to investigate the rate of occurrence of urethral pain when using GentleCath™ Air catheters as a bladder emptying method.

In this multicentre observational study each subject will participate for 90 days. Women under the care of the participating investigator and receiving their first prescription of GentleCath Air catheter for urinary dysfunction due to neurological disorders will be approached for potential participation in the study.

The primary outcome will be the pain assessment score measured on a VAS (Visual Analog Scale) during insertion and removal of the GentleCath™ Air catheter in naive female patients with confirmed neurological pathway on D1, D3, D7, D14, D21, D28, D35, D45 and D90.

The secondary outcomes will be to assess the patients' satisfaction of self-catheterization (based on InCaSaQ score) at D45 and D90, to describe patient compliance on D45 and D90, to measure the post-voiding residue on inclusion on D45 and D90, to assess compliance with the self-catheterization throughout study duration, to describe the tolerance of the GentleCath™ Air catheter throughout study duration and to measure the overall satisfaction on Gentle Cath Air on D90.

ELIGIBILITY:
Inclusion Criteria:

* Naive women of any self-catheterization,
* aged 18 years old or over,
* having been diagnosed with vesico-sphincteric disorders of neurological origin (spinal cord injury, multiple sclerosis, parkinsonian syndromes, ponytail syndrome),
* requiring self-catheterization and having a prescription for a GentleCath™ Air catheter.

Exclusion Criteria:

* Current participation in another clinical research,
* Patients not able to complete questionnaires.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women under the care of the participating investigator and receiving their first prescription of GentleCath Air catheter for urinary dysfunction due to neurological disorders will be approached for potential participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 1
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 3
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 7
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 14
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 21
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 28
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 35
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 45
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.
Pain assessment score during the insertion and removal of the GentleCath™ Air urinary catheter in female patients with confirmed neurological pathway | Day 90
  The pain assessment score will be measured on a VAS (Visual Analog Scale). The scale has a minimum value of 0 and a maximum value of 10. A higher score indicates a worse outcome indicating greater levels of pain and discomfort.

SECONDARY OUTCOMES:
Assessment of patients' satisfaction of self-catheterisation | Day 45
  The pain assessment score will be based on InCaSaQ score
Assessment of patients' satisfaction of self-catheterisation | Day 90
  The pain assessment score will be based on InCaSaQ score
Patient compliance | Day 45
  The proportion of patients continuing the self-catheterisation with the GentleCath™ Air catheter
Patient compliance | Day 90
  The proportion of patients continuing the self-catheterisation with the GentleCath™ Air catheter
Measurement of the post-voiding residue on inclusion | Day 45
  Post-catheterisation residue measurement (volume in mL) by ultrasound
Measurement of the post-voiding residue on inclusion | Day 90
  Post-catheterisation residue measurement (volume in mL) by ultrasound
Assessment of compliance with the self-catheterization - number of catheterizations | Day 1
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self--catheterization - number of catheterizations | Day 3
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-cathetization - number of catheterizations | Day 7
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 14
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 21
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 28
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 35
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 45
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - number of catheterizations | Day 90
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The number of catheterisations per 24 hours will be measured.
Assessment of compliance with the self-catheterization - Volume measurements | Day 1
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 3
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 7
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 14
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 21
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 28
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 35
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 45
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Assessment of compliance with the self-catheterization - Volume measurements | Day 90
  Assessment will be performed through review of self-reported outcomes via a patient diary with a completed voiding calendar. The volume per catheterisation, the 24-hour diuresis, leakage of urine between catheterisation and circumstances of leakage occurrence will be measured (volume in mL).
Description of the tolerance of the GentleCath™ Air catheter | Through study completion, approximately 13 months
  The proportion and description of adverse events occurring throughout the study follow-up period will be monitored
Measurement of the overall satisfaction on Gentle Cath Air | Day 90
  Patients will be questioned on the use of the catheter, service and products linked to GentleCath™ Air

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Gamé, Principal Investigator — Département d'Urologie, Transplantation Rénale et Andrologie, CHU Rangueil